CLINICAL TRIAL: NCT04876547
Title: Are Cesarean Section and Appendectomy in Pregnancy and Puerperium Interrelated?
Acronym: APPENDECTOMY
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Banuhan, Assistant professor, Amasya University
Other Study IDs: AmasyaU
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Appendicitis Acute; Cesarean Wound Disruption With Postnatal Complication
MeSH Terms: conditions — Appendicitis | interventions — Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- In pregnancy: Appendectomy in pregnancy (n=12)
  Interventions: Procedure: appendectomy
- In postpartum: Appendectomy in postpartum first six week (n=20)
  Interventions: Procedure: appendectomy

INTERVENTIONS:
Procedure: appendectomy — appendectomy performance

SUMMARY:
It is not known whether appendectomy for acute appendicitis (AA) increases the Cesarean section (CS) rate and whether CS increases the likelihood of AA and appendectomy in the early puerperium. In this study, delivery type and delivery outcomes and appendectomy during pregnancy and puerperium were analyzed.

DETAILED DESCRIPTION:
This cross-sectional retrospective study was performed on 11513 women, delivered during 2015-2020. Inclusion criteria were patients submitted to appendectomy for AA during pregnancy and the first six weeks after delivery. Evaluating parameters were age, parity, gestational week at birth, delivery type, and babies' birth weight.

ELIGIBILITY:
Inclusion Criteria: Women aged 18-45 years submitted to appendectomy for acute appendicitis during pregnancy or within the first six weeks after delivery were included.

-

Exclusion Criteria: Cases with missing data were excluded.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Study Population: Pregnant women who attended prenatal follow-up and delivered from October 1, 2015, to October 1, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
delivery type | 5 years
  vaginal birth, cesarean section

SECONDARY OUTCOMES:
Newborn weight | 5 years
  kg

OTHER OUTCOMES:
Cesarean indications | 5 years
  Fetal distress, dystocia, breech position

CONTACTS AND LOCATIONS:
Overall Officials: Banuhan Şahin, Principal Investigator — Gynecology and Obstetrics
Locations (1):
- Banuhan Şahin, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No